CLINICAL TRIAL: NCT06073067
Title: Safety, Efficacy, and Mechanism of Pre-operative Spatially Fractionated GRID Radiation Therapy in Patients With Extremity Soft Tissue Sarcoma: A Pilot Study
Brief Title: GRID Therapy for Extremity Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Radiation Oncology Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2250-DCT
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Sarcoma
Keywords: extremity; radiation; GRID; surgery; preoperative
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fractionated grid radiation therapy (Experimental): Subjects with resectable extremity soft tissue sarcoma received neoadjuvant grid radiation therapy (GRID), followed by standard-of-care conventional radiotherapy (XRT) and tumor resection.
  Interventions: Radiation: GRID therapy

INTERVENTIONS:
Radiation: GRID therapy — GRID therapy delivers a high dose of radiation to small areas of tumor interleaved with areas that intentionally receive a low dose

SUMMARY:
Patients with extremity soft tissue sarcoma (STS) are at high risk of recurrence. Pre-operative radiotherapy is used to increase the safe removal of tumors and improve local control in these patients. Increasing the preoperative radiotherapy dose with standard techniques might lead to normal tissue toxicity and postoperative wound complications.

GRID radiation therapy is a technique that may increases radiation dose with minimal added toxicity. It is hypothesized that GRID radiation dose will improve tumor response without increasing post-operative wound complications. While GRID has been used in many patients, there have been few formal studies to evaluate the safety and efficacy of the technique. In this study, a single priming dose of GRID will be administered to subjects with high-risk extremity soft tissue sarcoma prior to standard radiotherapy and tumor resection to determine the safety and clinical efficacy of the GRID dose. This single-arm pilot study will assess the safety of spatially fractionated grid radiation therapy (GRID) on 20 subjects with resectable extremity soft tissue sarcoma, followed by standard-of-care conventional radiotherapy (XRT) and tumor resection.

ELIGIBILITY:
In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Inclusion Criteria:

1. Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information. Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
2. Age ≥ 18 years at the time of consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 - 2 (Karnofsky Performance Status equivalent of 50 - 100).
4. Histological or cytological evidence/confirmation of extremity soft tissue sarcoma as determined by core-needle biopsy or excision biopsy. If the diagnostic tissue is not available or sufficient to perform correlative studies, must be willing to provide the mandatory pre-treatment core-needle biopsy. In some cases of extremity STS, subjects undergo an attempted surgical resection for a presumed benign condition and the specimen reveals malignancy. Such subjects are allowed so long as a complete, oncologic, resection was not performed/attempted and there is ≥ 5 cm of the remaining primary tumor.

Exclusion Criteria:

Subjects meeting any of the exclusion criteria listed below at baseline will be excluded from the study.

1. Subjects who have received prior radiotherapy to the tumor site.
2. Subjects who have undergone complete tumor resection of the primary tumor or who have developed tumor recurrence after resection.
3. History of serious or non-healing wound, ulcer, or bone fracture in the treatment limb within the last 5 years.
4. History of clinically significant lymphedema in the treated limb.
5. History of lupus, scleroderma, Sjogren's syndrome, Ehlers-Danlos syndrome (any type), or other collagen vascular disease that may pose a relative contraindication, due to increased risk of skin or soft tissue toxicity, with radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or higher post-operative wound complications after GRID-3 months | 3 months
  Safety will be quantified as the incidence of Grade 2 or higher post-operative wound complications after GRID, the standard of care XRT, and surgery.
  Wound complications will be graded according to The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  CTCAE is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.

SECONDARY OUTCOMES:
The tumor specimen of the surgery | At the time of surgery (Approximately 17th week)
  The effect of GRID on tumor response will be measured using the tumor specimen of the surgery. The major pathological response (MPR) rate will be defined as the viable residual tumor in 10% or less of the resection specimen.
Grade 2 or higher post-operative wound complications after GRID-6 months | 3 months to 6 months
  Safety will be quantified as the incidence of Grade 2 or higher post-operative wound complications after GRID, the standard of care XRT, and surgery.
  Wound complications will be graded according to The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  CTCAE is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Long Term Safety | 6 months after completrion of radiotherapy
  Safety will be quantified as the incidence of Grade 2 or higher post-operative wound complications after GRID, the standard of care XRT, and surgery.
  Wound complications will be graded according to The NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  CTCAE is a descriptive terminology that can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
The comparative effect of GRID | At the time of surgery (Approximately 17th week after completion of radiotherapy)
  The comparative effect of GRID will be quantified using histopathologic substrates. Comparisons will be made between pre-treatment biopsies, biopsies taken from different dose regions of the tumor specimen following GRID, and samples of the surgically resected tumor. The viable tumor rate will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore K Yanagihara, MD. PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials